CLINICAL TRIAL: NCT00000857
Title: A Phase I, Double-Blind, Randomized, Placebo-Controlled Trial of Recombinant Human Interleukin-12 (rhIL-12) in HIV-Infected Subjects With Less Than 50 CD4+ T Cells and Subjects With 300-500 CD4+ T Cells
Brief Title: A Study to Evaluate the Effects of Interleukin-12 (rhIL-12) in HIV-Positive Patients With CD4 Cell Counts Less Than 50 Cells/mm3 or 300-500 Cells/mm3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 325; 11299 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Recombinant Proteins; T-Lymphocytes; Dose-Response Relationship, Drug; Mycobacterium avium Complex; CD4 Lymphocyte Count; Interleukin-12; Killer Cells, Natural; Th1 Cells; Interferon Type II
MeSH Terms: conditions — HIV Infections; Mycobacterium avium-intracellulare Infection | interventions — Interleukin-12

INTERVENTIONS:
Drug: Interleukin-12

SUMMARY:
The purpose of this study is to determine the tolerance and effectiveness of rhIL-12 in HIV-positive patients with CD4 cell counts less than 50 cells/mm3 versus 300-500 cells/mm3. This study will look at the ability of rhIL-12 to boost the immune system against HIV and HIV-associated bacterial infections in these patients.

IL-12 is found naturally in the body and rhIL-12 is the commercially produced version. IL-12 may enhance anti-HIV immune system activity by increasing the number of cells that fight infection. IL-12 may also increase the body's ability to fight bacterial infections such as Mycobacterium avium complex (MAC).

DETAILED DESCRIPTION:
IL-12 has a number of effects in vitro that could be relevant to HIV disease including promotion of TH1 cell development, enhancement of HIV-specific T cell responses in cells from subjects with AIDS, and, of particular relevance to MAC disease, increasing secretion of cytotoxic cytokines such as IFN-gamma from both T lymphocytes and NK cells.

Part A (36 patients with less than 50 CD4+ cells/mm3):

Patients are randomized within one of three sequential dose cohorts and receive either rhIL-12 or matching placebo by subcutaneous injection twice weekly for four weeks. Eligible patients will participate in only 1 of the 3 dosing cohorts. Dose escalation to a new cohort of patients in Part A will occur only if all 3 of the following occur:

(1) At least 9 patients in the rhIL-12 arm have been enrolled in the current dose group and have either been on study drug for at least 4 weeks (temporary discontinuation is allowed) or have permanently discontinued study drug due to a primary toxicity endpoint.

[(2) AS PER AMENDMENT 6/16/97: Fewer than 2 of the 12 patients receiving rhIL-12 at 30 or 100 ng/kg have had a primary toxicity endpoint.] (3) Adequate data from a Genetics Institute/Wyeth Ayerst-sponsored dose escalation trial have been obtained and analyzed to demonstrate the safety of the dose to be administered to the next cohort.

Note: If 3 or more patients in the rhIL-12 arm of a given dose in Part A experience a primary toxicity endpoint, then accrual and further drug administration will be discontinued.

[AS PER AMENDMENT 6/16/97: If a cohort has exactly two patients in the rhIL-12 arm that experience a primary toxicity endpoint, then the next cohort receives study drug at the same dose as the current cohort, but administered only once a week. If a cohort receiving study drug administered once a week has at least two subjects experience a primary toxicity endpoint, then further drug administration in Part A is stopped. Any cohort that receives study drug once a week is the last cohort in Part A; no further dose escalation is performed].

Part B (18 subjects with 300-500 CD4+ cells/mm3):

Patients are randomized to receive either the maximum tolerated dose (determined in Part A) of rhIL-12 or matching placebo subcutaneously twice a week for 4 weeks.

[AS PER AMENDMENT 01/29/99: Because of slow accrual for cohort 3 of Part A, concurrent enrollment will begin for Part B while cohort 3 of Part A is completed. There will be no further dose escalation in Part A. Part A will remain open to accrual until the final enrollee to Part B completes 4 weeks of study treatment. For Part B, 27 patients will be randomized with equal probability to one of two rhIL-12 doses or placebo. Semiweekly injections are given for 4 weeks.]

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Are 18-60 years old.
* Have a CD4 count less than 50 cells/mm3 or between 300-500 cells/mm3 within 30 days of study entry.
* Are expected to live at least 12 weeks.
* Agree to practice abstinence or use effective methods of birth control during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have a history of cytomegalovirus (CMV) end-organ disease.
* Have a history of invasive fungal disease, unless the condition has been stable for 2 months.
* Have a history of severe allergic reactions to IL-2 or IL-12.
* Have a history of heart problems, autoimmune or rheumatologic disease, gastrointestinal bleeding, or any condition that would keep you from completing the study.
* Have MAC-related symptoms (fever, weight loss, frequent diarrhea) for at least 2 months prior to study entry.
* Are enrolled in another experimental research treatment study.
* Abuse alcohol or drugs.
* Are pregnant or breast-feeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65
Dates: Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jacobson, Study Chair; Richard Pollard, Study Chair
Locations (16):
- United States (16):
  - UCLA CARE Center CRS, Los Angeles, California
  - USC CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsf Aids Crs, San Francisco, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Weiss Memorial Hosp., Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Jacobson MA, Spritzler J, Landay A, Chan E, Katzenstein D, Schock B, Fox L, Roe J, Kundu S, Pollard R; AACTG 325 Protocol Team. A Phase I, placebo-controlled trial of multi-dose recombinant human interleukin-12 in patients with HIV infection. AIDS. 2002 May 24;16(8):1147-54. doi: 10.1097/00002030-200205240-00008. PMID 12004273